## Supplement to the Statistical Analysis Plan

Over the past five years, the Swedish maternal healthcare system has undergone significant changes in guidelines and practices. For example, national recommendations for induction of labour due to prolonged pregnancy have been moved from gestational week 42+0 to week 41+0. Additionally, diagnostic criteria for gestational diabetes, gestational hypertension, and preeclampsia have also changed, resulting in more women receiving these diagnoses, which affects the management of their pregnancy and delivery. To obtain more reliable data, we have therefore chosen not to use a historical control group. Instead, the control group will consist of women born in Somalia who gave birth during the same time interval as the intervention was implemented, but who were registered at a midwifery clinic that did not recieve the Mindfetalness intervention. We believe this will lead to a more credible analysis.